CLINICAL TRIAL: NCT04733482
Title: The Effects of Cosmetic Care on Body Image in Young Chinese Breast Cancer Patients Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhenqi Lu (Other)
Responsible Party: Sponsor-Investigator, Zhenqi Lu, Director of nursing department in Fudan University Shanghai Cancer Center, Fudan University
Organization: Fudan University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FNF201413
Record Dates: First submitted 2021-01-24; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Body Image
Keywords: body image; cosmetic care; psychosocial support; social avoidance and distress; young breast cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants in the control group received usual care during adjuvant chemotherapy. The usual care consisted of written information and verbal guidance on the adverse effects of chemotherapy and related psychological reactions.
- Cosmetic care group (Experimental): Participants in the intervention group received cosmetic care in combination with usual care. The cosmetic care was a 3-hour, free-of-charge beauty activity, including face moisturizing steps, make-up, wigs, and breast prostheses wearing. It was provided by professional cosmeticians at a cosmetic training base before the patients finished half of their chemotherapy cycle.
  Interventions: Behavioral: Cosmetic care

INTERVENTIONS:
Behavioral: Cosmetic care
  Arms: Cosmetic care group

SUMMARY:
This study aimed to explore the effects of cosmetic care on body image (BI), and social avoidance and distress (SAD) in young Chinese breast cancer patients, aged 18-40 years old, receiving adjuvant chemotherapy. This was a single-center, 2-arm quasi-experimental study. The control group received usual care, while cosmetic care was added to the intervention group. The primary outcomes were BI and SAD accompanying chemotherapy, and the secondary outcome was the appearance satisfaction.

DETAILED DESCRIPTION:
Background: The diagnosis and treatment of breast cancer may still bring severe psychological trauma to women. Cosmetic care is an effective measure to enhance patients' psychosocial functioning, which can help cancer patients cope with disfigurement-related adverse effects.

Objectives: This study aimed to explore the effects of cosmetic care on body image (BI), and social avoidance and distress (SAD) in young Chinese breast cancer patients, aged 18-40 years old, receiving adjuvant chemotherapy.

Study design: This was a prospective, 2-arm quasi-experimental study, comprising two groups: the controlled group and the interventional group. In order to avoid interference, the two groups of participants were recruited at different periods. The control group was recruited from Jan 2015 to Mar 2015, and the intervention group was recruited from January 2016 to September 2017. All participants came from the department of a breast surgery in Shanghai, China.

Control condition: Participants in the control group received usual care during adjuvant chemotherapy.

Intervention: Participants in the intervention group received cosmetic care in combination with usual care.

Ethical approval: Ethical approval of this study was obtained from the ethical committee of a cancer center in Shanghai. The approval number was 1403132-2. Informed consent was explained to the participants and the forms were signed by them.

Data analyses: The IBM SPSS 22.0 was used to analyze all the data.

ELIGIBILITY:
Inclusion Criteria:

* Primary breast cancer patients
* Aged 18-40 years old, who received surgery and adjuvant chemotherapy in our department
* No prior neoadjuvant chemotherapy
* Being available to communicate by the novel social application "Wechat"

Exclusion Criteria:

* Diagnosis of psychiatric or intellectual impairment
* Having a history of neoadjuvant therapy
* Having distant metastasis
* ECOG<2

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2015-01-03 (Actual); Primary Completion 2015-09-10 (Actual); Study Completion 2017-09-10 (Actual)

PRIMARY OUTCOMES:
Body image scale | Change from baseline to half of the cycle of chemotherapy and the end of cycle of chemotherapy (each cycle is 21 days, and there were 4-6 cycles totally).
  Body image (BI) was assessed using the body image scale. It is a 10-item self-assessment scale, measuring cancer patients' perception of their appearance. The minimum and maximum values of the scale are 0 and 30. A higher score signifies a worse BI.
Social avoidance and distress scale | Change from baseline to half of the cycle of chemotherapy and the end of cycle of chemotherapy (each cycle is 21 days, and there were 4-6 cycles totally.)
  Social avoidance and distress (SAD) was assessed using social avoidance and distress scale, which contains 28 items. The total score in the scale ranges from 0 to 28. A higher score means greater SAD.

SECONDARY OUTCOMES:
Appearance satisfaction questionnaire | The end of cycle of chemotherapy (each cycle is 21 days, and there were 4-6 cycles totally.).
  The appearance satisfaction questionnaire was designed by the researchers of this study, and aimed to assess whether the several body image- related side effects of treatments would affect patients' appearance satisfaction. It involved six aspects: hair loss, facial skin pigmentation, acne skin, breast loss, weight gain, and fatigue. The answers included either a "Yes" or a "No." The description of each item was used percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Shengqun Hou, Master, Principal Investigator — Fudan University; Zhenqi Lu, Master, Study Chair — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China